CLINICAL TRIAL: NCT05530096
Title: Detect and Profile Multiple Myeloma Measurable Residual Disease (MRD )Prognostics for Monitoring Post-transplant Multiple Myeloma (MM) Patients Receiving Maintenance Therapy.
Brief Title: Telo Genomics Technology to Detect & Profile Multiple Myeloma MRD
Acronym: TELO - DMRD
Status: Recruiting | Type: Observational
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Rayan Kaedbey, Principal Investigator, Sir Mortimer B. Davis - Jewish General Hospital
Other Study IDs: Telo Genomics Study
Record Dates: First submitted 2022-08-31; First posted 2022-09-07 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- MRD level group: Participants will be defined as diagnosed with multiple myeloma
  Interventions: Diagnostic Test: Standard of care

INTERVENTIONS:
Diagnostic Test: Standard of care — Participants will not receive any intervention in this study. Participants will receive standard of care therapy

SUMMARY:
The purpose :

Detect and profile Multiple myeloma Measurable Residual Disease(MRD) prognostics for monitoring post-transplant Multiple Myeloma (MM) Patients receiving maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed MM diagnosis
* Transplant eligible patients in a first remission
* Known MRD level detected by ClonoSeq (other IMWG recognized methodologies can be also employed)
* Availability of deidentified patient's demographic and clinical follow up data
* Receiving standard of care treatment
* Able to provide informed consent

Exclusion Criteria:

* Failure to meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant having confirmed Multiple Myeloma diagnosis will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
To validate the sensitivity of Telo Genomics assay (measurement tool) to detect MRD (measurement expressed in the number of plasma cells per 100000 cells) and establish the clinical utility of TELO - DMRD for MRD enumeration | Approximately 5 years
  Assess the possibility to perform TELO-DMRD on bone marrow aspirate samples vs peripheral blood
  Validate TELO-DMRD results with ClonoSeq, as an IMWG recognized MRD assessment method (other IMWG recognized methodologies can be also employed)
To assess the utility of TeloView® technology genomic profiling (measurement tool) to stratify post-transplant MM patients into relapse risk groups (dichotomous measure of high or low) by analyzing the residual MRD plasma cells | Approximately 5 years
  o A longitudinal study including transplant eligible patients. Patients to be followed for 6 time points over 24 months at: At point of diagnosis (marrow aspirate & peripheral blood), 4m post induction (peripheral blood), 3m Post-transplant (peripheral blood), at 12m Post-transplant (peripheral blood), 18m Post-transplant (peripheral blood) & 24m Post-transplant (peripheral blood), and at point of relapse for patients who will relapse during the follow up time (marrow aspirate & peripheral blood). Of note, an additional marrow aspirate may be performed if the patient agrees at the time they attain a complete remission, to confirm this status

CONTACTS AND LOCATIONS:
Overall Officials: Rayan Kaedbey, Principal Investigator — Sir Mortimer B. Davis - Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada